CLINICAL TRIAL: NCT04234204
Title: A Phase 3, Randomized, Placebo-controlled, 12-week Double-blind Study, Followed by a Non-Controlled Extension Treatment Period, to Assess the Efficacy and Safety of Fezolinetant in Women in Asia Suffering From Moderate to Severe Vasomotor Symptoms (Hot Flashes) Associated With Menopause
Brief Title: A Study to Find Out if Fezolinetant Helps Reduce Moderate to Severe Hot Flashes in Women in Asia Going Through Menopause
Acronym: Moonlight 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2693-CL-0305; CTR20200360 (Registry Identifier: ChinaDrugTrials.org.cn)
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Hot Flashes
Keywords: ESN364; menopause; fezolinetant; vasomotor symptoms
MeSH Terms: conditions — Hot Flashes | interventions — fezolinetant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fezolinetant group (Experimental): Participants will receive fezolinetant once daily for 24 weeks.
  Interventions: Drug: Fezolinetant
- Placebo group (Placebo Comparator): Participants will receive matching placebo for 12 weeks, and then receive fezolinetant for 12 weeks once daily.
  Interventions: Drug: Fezolinetant; Drug: Placebo

INTERVENTIONS:
Drug: Fezolinetant — Oral
  Other Names: ESN364
Drug: Placebo — Oral
  Arms: Placebo group

SUMMARY:
This study is for women in menopause with moderate to severe hot flashes. Menopause, a normal part of aging, is the time of a woman's last period. Hot flashes can interrupt a woman's daily life.

The study treatments are fezolinetant (1 tablet) once a day or placebo (1 tablet) once a day. (Placebo is a dummy treatment that looks like medicine but does not have any medicine in it.) The study will compare fezolinetant and placebo after 4 and 12 weeks of dosing. The study will see if fezolinetant reduces the number of hot flashes. And the study will see if fezolinetant reduces the severity of the hot flashes.

Women in the study will receive an electronic handheld device at the first study visit. (It is similar to a smart phone.) Each day of the study, study participants will use this to record their hot flashes. Their record for the 10 days before the start of study treatment will be checked. They can remain in the study if their record shows 7 or 8 moderate to severe hot flashes per day (50 or more per week).

Next, they will be picked for 1 of the 2 study treatments (fezolinetant or placebo) by chance alone. It is like flipping a coin.

The study participants will take study treatment for 24 weeks. The first 12 weeks of study treatment are "double-blinded." That means that the study participants and the study doctors do not know who takes which of the study treatments (fezolinetant or placebo) during that time. The last 12 weeks of study treatment are "noncontrolled." That means that each study participant and the study doctors know which study treatment that study participant takes during that time. Women who take fezolinetant during the first 12 weeks will continue to take fezolinetant. Women who take placebo during the first 12 weeks will start taking fezolinetant.

At weeks 2, 4, 8, 12, 14, 16, 20 and 24, the study participants will go to the hospital or clinic for a check-up. They will be asked about medications, side effects and how they feel. Other checks will include physical exam and vital signs (heart rate, temperature and blood pressure). Blood and urine will be collected for laboratory tests. Study participants will complete questionnaires that are about how hot flashes affect their daily life. Study participants who still have their uterus will have the following 2 tests done at the first and last study visits if they meet the criteria. One of the 2 tests is endometrial biopsy.

This test involves removing a small amount of tissue from the inside lining of the uterus. The tissue is then checked under a microscope. The other test is transvaginal ultrasound. This test uses sound waves to create pictures of the organs in the pelvis. The sound waves are transmitted by a probe (transducer), which is placed inside the vagina. Study participants may have a screening mammogram done at the first and/or last study visit. A mammogram is an x-ray picture of the breasts used to screen for breast cancer. Study participants who did not have this test done in the last 12 months will have it done at the first study visit. They will have it done at the last study visit if they are due for their screening mammogram and their own doctor agrees.

The last check-up at the hospital or clinic will be 3 weeks after the last dose of study treatment.

DETAILED DESCRIPTION:
This study will consist of a screening period and a 24-week treatment period. Safety follow up will occur 3 weeks after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a body mass index ≥16 kg/m^2 and ≤38 kg/m^2 (extremes included) at screening visit.
* Participant must be seeking treatment or relief for vasomotor symptoms (VMS) associated with menopause and confirmed as menopausal per 1 of the following criteria at the screening visit:

  * Spontaneous amenorrhea for ≥ 12 consecutive months
  * Spontaneous amenorrhea for ≥ 6 months with biochemical criteria of menopause (follicle stimulating hormone [FSH] > 40 IU/L); or
  * Having had bilateral oophorectomy ≥ 6 weeks prior to the screening visit (with or without hysterectomy)
  * FSH > 40 IU/L if participants received hysterectomy but still have ovary
* Within the 10 days prior to randomization, participant must have a minimum average of 7 to 8 moderate to severe HFs (VMS) per day, or 50 to 60 per week.
* Participant is in good general health as determined on the basis of medical history and general physical examination, including a bimanual clinical pelvic examination and clinical breast examination devoid of relevant clinical findings, performed at the screening visit; hematology and biochemistry parameters, pulse rate and/or blood pressure, and electrocardiogram (ECG) within the reference range for the population studied, or showing no clinically relevant deviations.
* Participant has documentation of a normal/negative or no clinically significant findings mammogram (or echo) (e.g. < BI-RADS class 4; obtained at screening or within the prior 12 months of study enrollment). Appropriate documentation includes a written report or an electronic report indicating normal/negative or no clinically significant mammographic findings.
* Participant is willing to undergo a transvaginal ultrasound (TVU) to evaluate the uterus and ovaries at screening and week 24 (end-of-treatment), and for participants who are withdrawn from the study prior to completion, a TVU at the early discontinuation (ED) visit. This is not required for participants who have had a partial (supra-cervical) or full hysterectomy.
* Participant is willing to undergo an endometrial biopsy at screening, and at week 24 (end of treatment) or early discontinuation (ED) visit if endometrial thickness >4mm indicated by TVU; and participant is willing to undergo an endometrial biopsy at any time during the study in the case of uterine bleeding. This is not required for participants who have had a partial (supracervical) or full hysterectomy. A biopsy with insufficient material for evaluation, or unevaluable material, is acceptable provided the endometrial thickness is no greater than 8 mm.
* Participant has documentation of a normal or not clinically significant Pap test (or equivalent cervical cytology within the previous 12 months of study enrollment or at screening. This is not required for participants who have had a full hysterectomy.
* Participant has a negative urine pregnancy test at screening, this is not required for participants who have had a full hysterectomy.
* Participant has negative serology panel [i.e., negative hepatitis B surface antigen (HBsAg) and negative hepatitis C virus antibody (HCVAb) screens] at screening.
* Participant agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Participant uses a prohibited therapy (strong and moderate cytochrome P450 1A2 [CYP1A2] inhibitors, hormone replacement therapy [HRT], hormonal contraceptive or any treatment for VMS [prescription, over the counter, or herbal]) or is not willing to wash out and discontinue use of such drugs for the full duration of study conduct.
* Participant has known substance abuse or alcohol addiction within 6 months of screening.
* Participant has a history of a malignant tumor, except for non-metastatic basal cell carcinoma of the skin.
* Participant has uncontrolled hypertension, defined as systolic blood pressure ≥ 140 mmHg or diastolic blood pressure as ≥ 90 mmHg based on an average of 2 to 3 readings within the screening period. Participants with a medical history of hypertension who are well controlled may be enrolled. Participants who do not meet these criteria may, at the discretion of the investigator, be re-assessed after initiation or review of antihypertensive measures.
* Participant has a history of severe allergy, hypersensitivity, or intolerance to drugs in general, including the study drug and any of its excipients.
* For Participants with a uterus: Participant has an unacceptable result from the TVU assessment at screening, i.e. full length of endometrial cavity cannot be visualized or presence of a clinically significant finding.
* For Participants with a uterus and endometrial thickness >4mm indicated by TVU: Participant has an endometrial biopsy confirming presence of disordered proliferative endometrium, endometrial hyperplasia, endometrial cancer, or other clinically significant at screening. A biopsy with insufficient material for evaluation, or unevaluable material is acceptable provided the endometrial thickness is no greater than 8 mm.
* Participant has a history within the last 6 months of undiagnosed uterine bleeding.
* Participant has a history of seizures or other convulsive disorders.
* Participant has a medical condition or chronic disease (including history of neurological [including cognitive], hepatic, renal, cardiovascular, gastrointestinal, pulmonary [e.g., moderate asthma], endocrine, or gynecological disease) or malignancy that could confound interpretation of the study outcome.
* Participant has active liver disease, jaundice, elevated liver aminotransferases (alanine aminotransferase [ALT] or aspartate aminotransferase [AST]), elevated total or direct bilirubin, elevated INR or elevated alkaline phosphatase (ALP). Patients with mildly elevated ALT or AST up to < 1.5 × the upper limit of normal (ULN) can be enrolled if total and direct bilirubin are normal. Patients with mildly elevated ALP (up to < 1.5 × ULN) can be enrolled if cholestatic liver disease is excluded and no cause other than fatty liver is diagnosed. Patients with Gilbert's syndrome with elevated total bilirubin may be enrolled as long as hemolysis is ruled out (i.e. direct bilirubin, hemoglobin and reticulocytes are normal).
* Participant has creatinine > 1.5 × ULN; or estimated glomerular filtration rate (eGFR) using the Modification of Diet in Renal Disease formula ≤ 59 mL/min/1.73 m^2 at screening.
* Participant has a positive result for human immunodeficiency virus (HIV) at screening.
* Participant has a history of suicide attempt or suicidal behavior within the last 12 months or has suicidal ideation within the last 12 months (a response of "yes" to question 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale [C-SSRS]), or who is at significant risk to commit suicide at screening and at visit 2.
* Participant has previously been enrolled in a clinical trial with fezolinetant.
* Participant has received investigational study drug within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Participant is unable or unwilling to complete the study procedures.
* Participant has any condition which makes the subject unsuitable for study participation.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in the frequency of moderate to severe vasomotor symptoms (VMS) | Baseline to Week 4
  Frequency of moderate or severe VMS events will be calculated as the sum of moderate or severe VMS events per day.
Mean change from baseline in the frequency of moderate to severe VMS | Baseline to Week 12
  Frequency of moderate or severe VMS events will be calculated as the sum of moderate or severe VMS events per day.
Mean change from baseline in the severity of moderate to severe VMS | Baseline to Week 4
  The severity of VMS will be calculated using a weighted average of VMS events.
Mean change from baseline in the severity of moderate to severe VMS | Baseline to Week 12
  The severity of VMS will be calculated using a weighted average of VMS events.

SECONDARY OUTCOMES:
Mean change from baseline to each week in the frequency of moderate and severe VMS | Baseline to Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 11, 12
  Frequency of moderate or severe VMS events will be calculated as the sum of moderate or severe VMS events per day.
Mean change from baseline to each week in the severity of moderate and severe VMS | Baseline to Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 11, 12
  The severity of VMS will be calculated using a weighted average of VMS events.
Mean percent reduction from baseline to each week in the frequency of moderate and severe VMS | Baseline to Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 11, 12
  Frequency of moderate or severe VMS events will be calculated as the sum of moderate or severe VMS events per day.
Percent reduction ≥50% from baseline to each week in the frequency of moderate and severe VMS | Baseline to Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 11, 12
  Frequency of moderate or severe VMS events will be calculated as the sum of moderate or severe VMS events per day. Ratio of the participants with ≥50% reduction in frequency will be reported.
Percent reduction at 100% from baseline to each week in the frequency of moderate and severe VMS | Baseline to Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 11, 12
  Frequency of moderate or severe VMS events will be calculated as the sum of moderate or severe VMS events per day. Ratio of the participants with ≥ 100% reduction in frequency will be reported.
Mean change from baseline in the frequency of moderate to severe VMS | Baseline to Week 24
  Frequency of moderate or severe VMS events will be calculated as the sum of moderate or severe VMS events per day.
Mean change from baseline in the severity of moderate to severe VMS | Baseline to Week 24
  The severity of VMS will be calculated using a weighted average of VMS events.
Number of Participants With Adverse Events | Up to 27 Weeks
  An adverse event (AE) is any untoward medical occurrence in a participant administered a study drug, and which does not necessarily have to have a causal relationship with this treatment.
Number of Participants With Adverse Events Based on Severity | Up to 27 Weeks
  An AE is any untoward medical occurrence in a participant administered a study drug, and which does not necessarily have to have a causal relationship with this treatment.
Change From Baseline in Endometrial Thickness | Baseline and Week 24
  Endometrial thickness is a measure of how thick the lining of the uterus is. Endometrial thickness will be measured by transvaginal ultrasound (TVU).
Percentage of Participants With Endometrial Hyperplasia and/or Endometrial Cancer | Up to 24 Weeks
  Endometrial hyperplasia is thickening of the lining of the uterus. Endometrial cancer is cancer of the lining of the uterus.
Number of Participants With Vital Sign Abnormalities and/or Adverse Events | Up to 27 Weeks
  Number of participants with potentially clinically significant vital sign values will be reported.
Number of Participants With Electrocardiogram (ECG) Abnormalities and/or Adverse Events (AEs) | Up to 27 Weeks
  Number of participants with potentially clinically significant ECG values will be reported.
Number of Participants With Laboratory Value Abnormalities and/or Adverse Events (AEs) | Up to 27 Weeks
  Number of participants with potentially clinically significant laboratory values will be reported.
Change From Baseline in Bone Specific Alkaline Phosphatase (BSAP) | Baseline, Week 24 and Week 27
  Change from baseline in serum concentrations of BSAP will be reported.
Change From Baseline in Procollagen Type 1 Aminoterminal Propeptide (P1NP) | Baseline, Week 24 and Week27
  Change from baseline in serum concentrations of P1NP will be reported.
Change From Baseline in Carboxy-Terminal Telopeptide of Type I Collagen (CTX) | Baseline, Week 24 and Week 27
  Change from baseline in serum concentrations of CTX will be reported.
Pharmacokinetics (PK) of Fezolinetant in Plasma: Concentration | Week 4, Week 12, Week 16, Week 24
  Concentration will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of Fezolinetant Metabolite ES259564 in Plasma: Concentration | Week 4, Week 12, Week 16, Week 24
  Concentration will be recorded from the PK plasma samples collected.
Change from Baseline in Sex Hormones | Baseline, Week 4, Week 12, Week 24 and Week 27
  Change from baseline in serum concentration of sex hormones will be reported.
Change from Baseline in Sex Hormone-Binding Globulin (SHBG) | Baseline, Week 4, Week 12, Week 24 and Week 27
  Change from baseline in serum concentration of SHBG will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma China, Inc.
Locations (48):
- China (31):
  - Site CN86001, Beijing
  - Site CN86002, Beijing
  - Site CN86017, Beijing
  - Site CN86030, Beijing
  - Site CN86022, Changchun
  - Site CN86009, Changsha
  - Site CN86037, Chengdu
  - Site CN86006, Guangzhou
  - Site CN86019, Guangzhou
  - Site CN86042, Guangzhou
  - Site CN86043, Guangzhou
  - Site CN86018, Guiyang
  - Site CN86025, Hangzhou
  - Site CN86034, Hangzhou
  - Site CN86027, Kunming
  - Site CN86005, Liuchow
  - Site CN86004, Nanjing
  - Site CN86011, Nanjing
  - Site CN86035, Nanjing
  - Site CN86026, Nanning
  - Site CN86012, Shanghai
  - Site CN86021, Shenzhen
  - Site CN86007, Shijiazhuang
  - Site CN86023, Taiyuan
  - Site CN86031, Taiyuan
  - Site CN86015, Tianjin
  - Site CN86029, Tianjin
  - Site CN86008, Wuhan
  - Site CN86041, Yangzhou
  - Site CN86013, Yinchuan
  - Site CN86033, Zhongshan
- South Korea (9):
  - Site KR82013, Ansan-si
  - Site KR82005, Busan
  - Site KR82003, Seongnam-si
  - Site KR82011, Seongnam-si
  - Site KR82001, Seoul
  - Site KR82002, Seoul
  - Site KR82004, Seoul
  - Site KR82006, Seoul
  - Site KR82012, Seoul
- Taiwan (8):
  - Site TW88608, Kaohsiung City
  - Site TW88604, New Taipei City
  - Site TW88606, Taichung
  - Site TW88603, Tainan
  - Site TW88609, Tainan
  - Site TW88601, Taipei
  - Site TW88607, Taipei
  - Site TW88611, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as compounds terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Ruan X, Bai W, Ren M, Kim T, Lee JY, Chuang FC, Wang PH, He W, Ma X, Miyazaki K, Song N, Wang X, Yu Q. Efficacy and safety of fezolinetant for moderate to severe vasomotor symptoms associated with menopause among women in East Asia: a phase 3 randomized study (MOONLIGHT I). J Int Med Res. 2024 May;52(5):3000605241247684. doi: 10.1177/03000605241247684. PMID 38818888
- See also: Link Description: Link to plain language summary of the study on the Trial Results Summaries website. — https://www.trialsummaries.com/Study/StudyDetails?id=14544&tenant=MT_AST_9011